CLINICAL TRIAL: NCT05889871
Title: A Randomized, Controlled, Open-label, Phase III Clinical Trial of Adjuvant Intensive Therapy for HR+/ HER2-SNF4 Early Breast Cancer Based on SNF Molecular Classification
Brief Title: A Randomized, Controlled, Open-label Clinical Trial of Adjuvant Intensive Therapy for HR+/ HER2-SNF4 Early Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N050
Record Dates: First submitted 2023-05-23; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: HR+/HER2-breast Cancer
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard endocrine therapy plus Apatinib (Experimental): 5 to 10 years of endocrine therapy (e.g., aromatase inhibitors, tamoxifen, LHRH agonists, etc.) and 2 years of CDK4/6 inhibitors, depending on clinical indications. plus Apatinib, 250mg orally once a day;
  Interventions: Drug: Standard endocrine therapy plus Apatinib
- Standard endocrine therapy (Active Comparator): 5 to 10 years of endocrine therapy (e.g., aromatase inhibitors, tamoxifen, LHRH agonists, etc.) and 2 years of CDK4/6 inhibitors, depending on clinical indications.
  Interventions: Drug: Standard endocrine therapy plus Apatinib

INTERVENTIONS:
Drug: Standard endocrine therapy plus Apatinib — Standard endocrine therapy plus Apatinib

SUMMARY:
This is a randomized, controlled, open, phase III trial of adjuvant intensive therapy for early breast cancer with HR+/ HER2-SNF4 based on SNF molecular typing. A randomized, controlled, open Phase III study to explore the efficacy and safety of Apatinib combined with standard endocrine therapy in adjuvant intensive therapy for HR+/ HER2-SNF4 type early high-risk breast cancer.

DETAILED DESCRIPTION:
584 patients with lumofacial breast cancer (ER and PR positive, HER2 negative) who received surgery in the Breast Surgery Department of the Affiliated Cancer Hospital of Fudan University were previously collected. The main work was genome sequencing (514 cases of whole exon sequencing, 527 cases of OncoScan microarray), 573 cases of transcriptome sequencing, 228 cases of proteomics (TMT mass spectrometry), 384 cases of metabolomics (liquid chromatography), 439 cases of digital pathology, and partial paired single cell transcriptome sequencing. This group ranks as the largest Asian coelfacial breast cancer multiomics cohort to date. All patients could be divided into four categories by SNF algorithm fusion clustering, namely SNF1 (classical coelateral type), SNF2 (immune-mediated type), SNF3 (proliferative type) and SNF4 (receptor tyrosine kinase-driven type). Different types had unique multiomics and clinicopathological characteristics, which fully analyzed the molecular heterogeneity of coelateral type breast cancer.

This is a randomized, controlled, open, phase III trial of adjuvant intensive therapy for early breast cancer with HR+/ HER2-SNF4 based on SNF molecular typing. A randomized, controlled, open Phase III study to explore the efficacy and safety of Apatinib combined with standard endocrine therapy in adjuvant intensive therapy for HR+/ HER2-SNF4 type early high-risk breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years and ≤70 years;
2. Histologically confirmed HR+/HER2- invasive breast cancer (defined by immunohistochemical detection of ER > 10% positive tumor cells were defined as ER positive, PR > 10% positive tumor cells were defined as positive PR, and ER and/or PR were defined as positive HR. HER2 0-1+ or HER2 ++ but negative by FISH test, no amplification, defined as HER2 negative);
3. Definition of SNF4 subtype: SNF4 subtype confirmed by digital pathology of H&E sections;
4. High-risk early breast cancer, which was pathologically confirmed as HR+/HER2- and SNF4 subtypes; pT2-4N0-3M0;
5. Complete the adjuvant chemotherapy selected by the doctor;
6. No more than 16 months from surgery to randomization, and no more than 12 weeks after non-endocrine therapy;
7. The functions of major organs are basically normal, meeting the following conditions:

   1. The standard of blood routine examination shall meet: HB ≥90 g/L (no blood transfusion within 14 days); ANC ≥1.5×109 /L; PLT ≥75×109 /L;
   2. Biochemical examination shall meet the following standards: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3 x ULN; In case of liver metastasis, ALT and AST≤ 5×ULN; Serum Cr ≤1×ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
8. ECOG score 0 or 1;
9. Fertile female subjects are required to use a medically approved contraceptive for the duration of the study treatment and for at least 3 months after the last use of the study drug; The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. bilateral breast cancer;
2. A history of other malignancies, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
3. transfer of any part;
4. Pregnant or lactating women, women of childbearing age can not effectively contraceptive;
5. Patients participating in other clinical trials;
6. Severe organ dysfunction (heart, lung, liver and kidney); 50% (cardiac hypertrophy); Severe cardiovascular and cerebrovascular disease (e.g., unstable angina, chronic heart failure, myocardial infarction, or cerebrovascular accident) within 6 months before randomization; Diabetics with poor blood sugar control;
7. Patients with a history of gastrointestinal bleeding or a definite tendency to gastrointestinal bleeding within the past 6 months, such as esophageal varicose veins with bleeding risk, locally active ulcer lesions, stool occult blood ≥ (++), shall not be included in the group; If fecal occult blood (+), gastroscopy is required;
8. Abdominal fistula, gastrointestinal perforation, or abdominal abscess in the 28 days before the study;
9. Urine routine showed urine protein ≥++ or confirmed 24 hours urine protein quantity > 1.0g;
10. Patients with hypertension who cannot be reduced to the normal range after antihypertensive medication (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg).
11. Allergic constitution, or known allergic history of the drug components of the program;
12. Previous thyroid dysfunction;
13. Severe or uncontrolled infection;
14. Those who have a history of psychotropic drug abuse and cannot abstain or have a history of mental disorders; The researchers determined that the patients were not suitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 916 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year survival without invasive disease (iDFS) | 3 years
  3-year survival without invasive disease (iDFS)

SECONDARY OUTCOMES:
3-year distant disease free survival (DDFS) | 3 years
  3-year distant disease free survival (DDFS)
5-year overall survival (OS) | 5 years
  5-year overall survival (OS)
security | through study completion, an average of 1 year
  Incidence of treatment-emergent adverse events adverse events according to CTCAE 5.0
PRO (patient reported outcome) | 5 years
  Registration of differences in quality of life between the two groups in the study. EORTC QLQ-C30(scale range 0-100, a higher score indicating better quality of life) will be used for as quality of life measurement. The scores will be presented graphically in separate figures. Differences between the groups will be tested using t-test and analysis of covariance.

IPD SHARING:
Plan to Share IPD: No